CLINICAL TRIAL: NCT00365885
Title: Showing Health Information Value in a Community Network
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00006833; R01HS015057 (AHRQ)
Record Dates: First submitted 2006-08-16; First posted 2006-08-18 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2012-12

CONDITIONS: Clinical Decision Support; Medical Informatics Interventions; Population Health Management; Quality of Healthcare
Keywords: Medical Informatics; Decision Support Systems, Clinical; Community Health Services; Costs and Cost analysis

STUDY DESIGN:
Who Masked: Participant

ARMS (6):
- 1 (Experimental): electronic mail notifications to care managers about sentinel health events
  Interventions: Other: Computer-based clinical decision support.
- 2 (Experimental): feedback reports with notifications to clinic managers about sentinel health events
  Interventions: Other: Computer-based clinical decision support.
- 3 (Experimental): letters to patients with notifications about sentinel health events
  Interventions: Other: Computer-based clinical decision support.
- 4 (No Intervention): electronic mail notifications to care managers about sentinel health events -- generated but withheld
- 5 (No Intervention): feedback reports with notifications to clinic managers about sentinel health events -- generated but withheld
- 6 (No Intervention): letters to patients with notifications about sentinel health events -- generated but withheld

INTERVENTIONS:
Other: Computer-based clinical decision support. — computer decision support system that generates notifications about sentinel health events and communicates this information via electronic mail to care managers, feedback reports to clinical managers, and letters to patients
  Other Names: Decision support engine is called SEBASTIAN
  Arms: 1; 2; 3

SUMMARY:
The purpose of this study is to determine the value of shared health information on care quality and costs when this information is used to notify care providers about concerning health events for patients cared for by a community-based network of providers.

DETAILED DESCRIPTION:
Project Abstract This three-year project will assess the costs and benefits of health information technology (HIT) in an established community-wide network of academic, private and public healthcare facilities created to share clinical information for the purpose of population-based care management of over 16,000 Medicaid beneficiaries in Durham County, North Carolina. The area of interest for this project is the impact of information-driven interventions on care quality, patient safety and healthcare costs across the diverse stakeholders participating in this collaborative partnership. In order to asses HIT value rigorously in the context of a production information system that is under continual development, we propose to conduct a randomized controlled trial. Specifically, we will randomly assign patients by family unit to either a control group or to an intervention group in which they will initially receive one of 3 information-driven interventions. The interventions include clinical alerts sent to care providers, performance feedback reports presented to clinic managers, and care reminders sent directly to patients. The content of the interventions will address "concerning" events (e.g., an emergency room encounter for asthma) and care deficiencies (e.g., delinquency on biannual mammogram) identified from the composite set of clinical data in our information system. To assess the benefits and burdens of the interventions, combinations of the 3 interventions will be sequentially introduced into the study groups over the course of the project. The analysis will compare groups receiving various combinations of interventions as well as those receiving no interventions. At baseline and at six-month intervals throughout the course of the study, we will measure emergency department encounter rates, hospitalization rates, HEDIS (Healthcare Effectiveness Data and Information Set) scores, missed appointment rates, glycated hemoglobin levels in diabetics, and patient satisfaction. Our assessment will look at the societal value of HIT as well as the value for individual stakeholders including patients, providers, payers, purchasers and policy makers. From these measures, we will assess the costs and benefits of this community-wide effort to promote interoperability of clinical data exchange in order to increase the understanding of HIT value in a community setting. In our preliminary studies, we have observed a statistically significant 3-fold reduction in repeat ED (Emergency Department) encounter rates using email alerts alone. The approach used in this project is able to be generalized across geographic areas and healthcare settings and can, therefore, serve to promote the dissemination of HIT to other communities.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in the Community Care of North Carolina Medicaid program in Durham County North Carolina

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20108 (Actual)
Dates: Start 2006-08; Primary Completion 2008-07 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Emergency department utilization rates and hospitalization rates | at 9 months after the intervention has been introduced and then at 6-month intervals as the intervention is sequentially enhanced.

SECONDARY OUTCOMES:
ED encounter rates for low severity conditions | at 9 months after the intervention has been introduced and then at 6-month intervals as the intervention is sequentially enhanced.
ED encounter rates for asthma | at 9 months after the intervention has been introduced and then at 6-month intervals as the intervention is sequentially enhanced.
ED encounter rates for diabetes | at 9 months after the intervention has been introduced and then at 6-month intervals as the intervention is sequentially enhanced.
Hospitalization rates | at 9 months after the intervention has been introduced and then at 6-month intervals as the intervention is sequentially enhanced.
Hospitalization rates for asthma (also PQI) | at 9 months after the intervention has been introduced and then at 6-month intervals as the intervention is sequentially enhanced.
Hospitalization rates for diabetes (also PQI) | at 9 months after the intervention has been introduced and then at 6-month intervals as the intervention is sequentially enhanced.
Glycemic control (hemoglobin A1c) | at 9 months after the intervention has been introduced and then at 6-month intervals as the intervention is sequentially enhanced.
Medication contraindications | at 9 months after the intervention has been introduced and then at 6-month intervals as the intervention is sequentially enhanced.
HEDIS - Preventive services | at 9 months after the intervention has been introduced and then at 6-month intervals as the intervention is sequentially enhanced.
HEDIS - # WCC visits | at 9 months after the intervention has been introduced and then at 6-month intervals as the intervention is sequentially enhanced.
AHRQ Prevention Quality Indicators | at 9 months after the intervention has been introduced and then at 6-month intervals as the intervention is sequentially enhanced.
HEDIS - Asthma and diabetes | at 9 months after the intervention has been introduced and then at 6-month intervals as the intervention is sequentially enhanced.
# of messages triggered for health risks | at 9 months after the intervention has been introduced and then at 6-month intervals as the intervention is sequentially enhanced.
# of messages triggered for barriers to care | at 9 months after the intervention has been introduced and then at 6-month intervals as the intervention is sequentially enhanced.
Missed appointment rates | at 9 months after the intervention has been introduced and then at 6-month intervals as the intervention is sequentially enhanced.
Primary care appointment rates | at 9 months after the intervention has been introduced and then at 6-month intervals as the intervention is sequentially enhanced.
F/U rates post-partum | at 9 months after the intervention has been introduced and then at 6-month intervals as the intervention is sequentially enhanced.
Patient satisfaction instruments (CHAPS) | at 6 to 9 months after the intervention has been introduced and then at 3 to 6-month intervals as the intervention is sequentially enhanced.
EuroQoL | at 6 to 9 months after the intervention has been introduced and then at 3 to 6-month intervals as the intervention is sequentially enhanced.
Provider opinion surveys | At conclusion of study
Costs of ED utilization for all causes | at 9 months after the intervention has been introduced and then at 6-month intervals as the intervention is sequentially enhanced.
Costs of ED use for asthma | at 9 months after the intervention has been introduced and then at 6-month intervals as the intervention is sequentially enhanced.
Costs of ED use for diabetes | at 9 months after the intervention has been introduced and then at 6-month intervals as the intervention is sequentially enhanced.
Costs of ED use for low severity visits | at 9 months after the intervention has been introduced and then at 6-month intervals as the intervention is sequentially enhanced.
Hospitalization costs for all causes | at 9 months after the intervention has been introduced and then at 6-month intervals as the intervention is sequentially enhanced.
Hospitalization costs for asthma | at 9 months after the intervention has been introduced and then at 6-month intervals as the intervention is sequentially enhanced.
Hospitalization costs for diabetes | at 9 months after the intervention has been introduced and then at 6-month intervals as the intervention is sequentially enhanced.
Reimbursement for labs+other ancillary services | at 9 months after the intervention has been introduced and then at 6-month intervals as the intervention is sequentially enhanced.
Primary care reimbursement | at 9 months after the intervention has been introduced and then at 6-month intervals as the intervention is sequentially enhanced.
ED rates for recurrent ED encounters | at 9 months after the intervention has been introduced and then at 6-month intervals as the intervention is sequentially enhanced.

CONTACTS AND LOCATIONS:
Overall Officials: David F Lobach, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Eisenstein EL, Anstrom KJ, Macri JM, Crosslin DR, Johnson FS, Kawamoto K, Lobach DF. Assessing the potential economic value of health information technology interventions in a community-based health network. AMIA Annu Symp Proc. 2005;2005:221-5. PMID 16779034